CLINICAL TRIAL: NCT02492724
Title: Activ C Disc Prosthesis European Multi-Center Clinical Investigation
Brief Title: Activ C European Multicenter Study
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-0707
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Intervertebral Disc Replacement; Degenerative Disc Disease
Keywords: cervical spine; total disc replacement (cTDR); degenerative disc disease; activ® C; clinical outcome; long-term results; NDI; VAS; heterotopic ossification (HO); range of motion (ROM); adjacent segment degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration; Ossification, Heterotopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients are candidates for single-level Artificial Disc Replacement between C3 and C7 who suffer from cervical symptomatic degenerative disc disease. A maximum of 200 cases will be enrolled into the study. An 18-month recruitment period is planned with a 4-year postoperative follow-up period for each subject. Thus, it is anticipated that the study will require a minimum of 5.5 years. Patients will be assessed preoperatively, intraoperatively, prior to discharge and again at 6 weeks, 6 months, 1 year, 2 years and 4 years postoperatively from the date of surgery.

DETAILED DESCRIPTION:
The activ C Disc Prosthesis pursues the goal of restoring the disc function, the geometry and motion of the cervical disc. Its concept is based on a ball and socket joint, anchored between adjacent vertebral bodies. The modular prosthesis comprises the following elements: an inferior CoCr plate component anchored in the endplate of the caudal vertebral body. The UHMWPE inlay is securely fixed in this inferior component. The second element is the superior CoCr component, which is anchored in the end plate of the cranial vertebral body. It forms a ball joint with the inlay of the inferior plate component.

The activ C product range enables reconstruction of various disc heights as well as adaptation to the end plate sizes. Secure primary anchorage of the prosthesis to the vertebral bodies is achieved by convexly shaped superior end pla tes and fixation means (spikes and grooves on the superior end plate, a small keel on the inferior end plate), whereas secondary stability is facilitated by an osseointegrative Plasmapore® coating.

The objective of the study is to collect outcome information on the Activ® C Disc Prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic single-level cervical degenerative disc disease with neck and/or arm
* pain and/or neurological deficit, confirmed by MR scan
* Single-level surgery and single-level implantation of prosthesis between C3 and C7
* Age between 18 - 65 years at the time of surgery
* Pre-operative disc space height of the segment to be operated of at least 3mm
* Unsuccessful adequate conservative treatment
* Patient understands the conditions of the study and is willing and able to comply with the post-operative scheduled clinical and radiographic evaluations and the prescribed rehabilitation
* Patient signed Informed Consent

Exclusion Criteria:

* Major facet joint degeneration at the segment to be operated on
* Severe spondylosis at the segment to be operated on (bridging osteophytes, absence of motion (<2°))
* Pre-operative disc space height of the segment to be operated on of less than 3mm
* Major cervical segmental instability at the segment to be operated on (translation ≥3,5 mm and/or ≥11° of rotational difference to that of either adjacent level)
* Previous trauma to the segment to be operated on resulting in compression or bursting

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2007-02; Primary Completion 2009-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Clinical Outcome measured by the Neck Disability Index (NDI) | 4 years
  The primary endpoint of the study will be changes in the clinical outcome measured by the Neck Disability Index (NDI) as published by Vernon et. al.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) on severity of neck pain and arm pain (experienced in the pain-dominant arm) | 4 years
Visual Analogue Scale (VAS) on frequency of neck pain and arm pain (experienced in the pain-dominant arm) | 4 years
Adjacent segment degeneration | 4 years
Postoperative angular motion on flexion/extension radiographs in the replaced segment | 4 years
Complication rates (device related and non-device related) | 4 years
Overall success rate | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Petr Suchomel, MD PhD, Principal Investigator — Neurocentre, Regional Hospital Liberec, Liberec, Czech Republic
Locations (10):
- Czechia (3):
  - Regional Hospital Liberec, Liberec
  - Faculty Hospital Motol Prague, Prague
  - University Hospital Motol, Prague
- Helsinki University Central Hospital, Helsinki, Finland
- Germany (4):
  - Charité Berlin, Berlin
  - Berufsgenossenschaftliche Kliniken Bergmannstrost, Halle
  - Katholisches Klinikum Koblenz, Koblenz
  - Universität Rostock, Abteilung Neurochirurgie, Rostock
- Neurosurgery at Instituti Fisioterapici Ospitalieri IFO, Rome, Italy
- Warrington District General Hospital, Warrington, United Kingdom

REFERENCES:
- [Result] Suchomel P, Jurak L, Antinheimo J, Pohjola J, Stulik J, Meisel HJ, Cabraja M, Woiciechowsky C, Bruchmann B, Shackleford I, Arregui R, Sola S. Does sagittal position of the CTDR-related centre of rotation influence functional outcome? Prospective 2-year follow-up analysis. Eur Spine J. 2014 May;23(5):1124-34. doi: 10.1007/s00586-014-3223-0. Epub 2014 Feb 20. PMID 24554334
- [Derived] Meisel HJ, Jurak L, Antinheimo J, Arregui R, Bruchmann B, Cabraja M, Caroli F, Kroppenstedt S, Kryl J, Pohjola J, Shackleford I, Sola S, Stosberg P, Stulik J, Woiciechowsky C, Suchomel P. Four-year results of a prospective single-arm study on 200 semi-constrained total cervical disc prostheses: clinical and radiographic outcome. J Neurosurg Spine. 2016 Nov;25(5):556-565. doi: 10.3171/2016.3.SPINE15810. Epub 2016 Jun 3. PMID 27258476